CLINICAL TRIAL: NCT02982499
Title: Biomechanics of Optic Neuropathy
Status: Terminated | Type: Observational
Why Stopped: Principal investigator's decision due to lack of resources
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Byron Lam, Professor, University of Miami
Other Study IDs: 20160376
Record Dates: First submitted 2016-08-28; First posted 2016-12-05 (Estimated); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Optic Neuropathy
Keywords: glaucoma; Leber optic neuropathy; anterior ischemic optic neuropathy
MeSH Terms: conditions — Optic Nerve Diseases; Glaucoma; Optic Atrophy, Hereditary, Leber; Optic Neuropathy, Ischemic | interventions — Magnetic Resonance Imaging; Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- control group: Healthy participants will receive a one-time assessment of quantitative Magnetic Resonance Imaging (MRI) and spectrum domain optical coherence tomography (OCT).
  Interventions: Device: magnetic resonance image (MRI); Device: Optical Coherence Tomography (OCT)
- optic neuropathy group: Participants with optic neuropathy will receive a one-time assessment of quantitative Magnetic Resonance Imaging (MRI) and spectrum domain optical coherence tomography (OCT).
  Interventions: Device: magnetic resonance image (MRI); Device: Optical Coherence Tomography (OCT)

INTERVENTIONS:
Device: magnetic resonance image (MRI) — Radiographic imaging that takes about 30-45 minutes
Device: Optical Coherence Tomography (OCT) — Images taken from the back of the eye (retina)

SUMMARY:
The participant is being asked to be a subject in this research study because the participant may have a disorder that can cause optic nerve damage and impairment of his/her visual function which is called optic neuropathies (ON). Optic neuropathy refers to damage to the optic nerve (a "cable" connecting the eyes and the brain to transmit the visual signals) due to any cause.In this study, the investigator is using magnetic resonance imaging (MRI) and ophthalmic measures such as optic coherent tomography(OCT), which are non-invasive imaging tests to measure the changes in eye globe shape ,the flow of blood and brain fluid. It is hoped that this study will provide new knowledge that may allow the investigator to better understand the cause of symptoms associated with optic neuropathy and ways to better monitor what is happening.

ELIGIBILITY:
Inclusion Criteria :

* 18 years old and on
* Patients with optic neuropathy(10) and age controlled healthy subjects(10)

Exclusion Criteria :

* For patients: Subjects with history of neurological or ocular disease other than optic neuropathy and refractory error.
* For healthy control group: History of systemic disease except hypertension.
* Pregnant women and prisoners will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Case group: Patients with optic neuropathy who are 18 years or older Control group: age-matched healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-03-26 (Actual); Study Completion 2018-03-26 (Actual)

PRIMARY OUTCOMES:
Globe deformation | day 1
  Three measures of globe deformation are calculated by using the distance map: 1) optic nerve cupping(ONC), depicting the extent of the nerve head cupping; 2) posterior scleral bowing, depicting the degree of displacement of the posterior wall, and 3) maximal deformation (MD), depicting the combined deformation due to the displacement and the nerve cupping.

SECONDARY OUTCOMES:
intracranial pressure | Day 1
  Intracranial pressure will be measured using non invasive MRI.
Corneal thickness | Day 1
  Corneal thickness will be measured by corneal pachymetry. After anesthetic numbing drop is placed on the eye, blunt probe will briefly touch the participant's eye to obtain the measurement.
Visual field defect | Day 1
  Humphrey Field Analyzer II will be used to acquire the Mean deviation(MD).

CONTACTS AND LOCATIONS:
Overall Officials: Byron R Lam, MD, Principal Investigator — University of Miami
Locations (1):
- Bascom Palmer Eye Institute, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No